CLINICAL TRIAL: NCT00321204
Title: A Retrospective Study of the Role of Thiazolidinediones to Reduce the Incidence of Atrial Arrhythmias in Patients After Cardiac Surgery
Brief Title: A Retrospective Study of the Role of Thiazolidinediones to Reduce the Incidence of Atrial Arrhythmias
Status: Terminated | Type: Observational
Why Stopped: Terminated: We are no longer recruiting.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Samuel C. Dudley, Jr., Principal Investigator, Emory University
Other Study IDs: IRB00002175; 1308-2005 (Other: Other)
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Atrial Flutter; Cardiac Surgery; Thiazolidinediones
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: TZD reducing the incidence of atrial arrhythmias

SUMMARY:
It is well known that abnormal heart beats from the top parts of the heart, atrial fibrillation (AF) and atrial flutter (Aflut), occur frequently after most types of cardiac surgeries. Postoperative AF and Aflut are associated with significant morbidity, longer hospital stay, and higher related costs. Currently therapies are marginally effective at preventing this abnormal heart beat. The incidence of abnormal heart beats after cardiac surgery seems to be a function of the amount of inflammation and oxidative stress induced. Our group and others have shown that atrial abnormal heart beats are associated with increased oxidative stress. Thiazolidinediones (TZDs) are medications used to treat diabetes. Beside their glucose lowering effects, TZDs are shown to exhibit anti-inflammatory and antioxidant properties. Therefore, we propose to retrospectively analyze the effect of pre-operative TZDs on the incidence of post-operative AF or Aflut. This study will involve retrospective chart reviews without further patient contact of all patients having undergone cardiac surgery in Emory University Hospital, Crawford Long Hospital, or the VA Medical Center from 2000 to 2005. This study is preparatory to a funding proposal for a prospective trial.

DETAILED DESCRIPTION:
1.0 Background

Cardiac surgery is associated with many perioperative complications, including supraventricular arrhythmias.(1-4) Atrial fibrillation occurs in 15 to 40% of patients after coronary artery bypass grafting (CABG) and up to 60% after CABG and valve repair. It can lead to significant complications such as stroke, prolonged hospitalizations, increasing mortality and morbidity.(1;5)

Post-operative atrial arrhythmias seem to be related to the degree of inflammation and oxidative stress induced during surgery.(2-4) Our group and others have shown that atrial arrhythmias are associated with increased oxidative stress.(6-10) Moreover, increased oxidative stress associated with angiotensin II-mediated NADPH oxidase activation leads to electrical abnormalities likely to propagate arrhythmias.(11;12)

Thiazolidinediones (TZDs) are antidiabetic agents that enhance insulin sensitivity through activating peroxisome proliferators-activated receptor (PPAR) gamma. Beside their glucose lowering effects, TZDs are shown to exhibit anti-inflammatory and antioxidant properties.(13-17)

2.0 Objectives

Based on the discussion above, we hypothesize that pre-operative use of TZDs will decrease post-operative AF or Aflut incidence. This study will be a retrospective cohort analysis of all patients that underwent elective cardiac surgeries between 2000-2005 at Emory University Hospital, Crawford Long Hospital, or the Atlanta Veterans Affairs Medical Center to evaluate the relationship of pre-operative TZD use to the incidence of post-operative atrial arrhythmias.. This study is undertaken in preparation for a funding proposal for a prospective trial.

3.0 Patient Selection

3.1 Eligibility criteria:

1. All patients that patients who underwent elective cardiac surgery in the Emory University Hospital, Crawford Long Hospital, or the VA Medical Center between 2000-2005.

3.2 Ineligibility criteria:

1. Emergent operations.
2. The presence of AF or Aflut at the time of surgery.
3. Patients without adequate documentation of atrial rhythm following surgery.
4. New York Heart Association (NYHA) class IV heart failure at the time of surgery.
5. Hyperthyroidism
6. Implanted devices for designed for active management of atrial arrhythmias by pacing or defibrillation
7. Known illicit drug use
8. Known ethanol abuse
9. Electrophysiological ablation for atrial tachycardia within 6 months of the operation.

4.0 Registration and randomization: none

5.0 Therapy: none

6.0 Pathology: none

7.0 Patient assessment: none

8.0 Data collection: Data will be collected from review of the patient's hospital charts, from telemetry recordings, and ECGs to document the presence or absence of AF or Aflut during the hospital admission for cardiac surgery. The presence or absence of atrial fibrillation will be diagnosed on the basis of an electrocardiographic recording and confirmed by a cardiologist. Demographic data collected will include: age, race, sex, body mass index, blood pressure, NYHA classification, Killip classification, and the history of previous myocardial infarction, hypertension, diabetes, smoking, alcohol use, antiarrhythmic drug use, presence and type of pacemaker if any, history of AF or Aflut, previous cardioversions, type of operation, and length of operation. Patients enrolled in this study will be given unique study numbers. No follow up data will be required from patients.

9.0 Statistical considerations: This study design is a retrospective chart review of a cohort of patients undergoing cardiac surgery to determine if there is an association between pre-operative TZD use and the incidence of post-operative atrial fibrillation or Aflut. The null hypothesis is that there is no association between the preoperative use of TZDs and postoperative AF and Aflut. Within the cohort, those patients with AF or Aflut will be compared to those without these atrial arrhythmias in the post-operative period. Baseline data for the two groups will be expressed as mean ± standard deviation for continuous variables, and frequencies for categorical variables. Differences in baseline characteristics between the groups will be examined by use of Fisher exact and Mann-Whitney tests for categorical and continuous variables, respectively. Quantification of any association between pre-operative TZD and the presence of atrial fibrillation will modeled by logistical regression analysis after adjusting for other variables that may affect arrhythmia frequency.

ELIGIBILITY:
Inclusion Criteria:

All patient who underwent elective cardiac Surgery in the Emory University Hospital, Crawford Long Hospital, or the Va Medical Center between 2000-2005.-

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2005-12; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel C. Dudley, Jr., MD, PhD, Principal Investigator — Veteran Administration Medical Center/Emory University
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Veteran Administration Medical Center, Decatur, Georgia